CLINICAL TRIAL: NCT06572930
Title: Assessment of the Role of Serum FSH Monitoring During Ovarian Stimulation and Identification of an Optimal Range for Expected Normal Responders
Brief Title: Serum FSH Monitoring for Identification of an Optimal Range During Ovarian Stimulation
Acronym: FSH
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2406-ABU-006-BA
Record Dates: First submitted 2024-08-08; First posted 2024-08-27 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Stimulation
Keywords: ovarian response; stimulation protocols; stimulation monitoring; follicular stimulating hormone
MeSH Terms: interventions — follitropin alfa; Gonadotropins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood tests, urine and follicular fluid for hormonal assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FSH Monitoring Group: Women undergoing ovarian stimulation will be given preselected constant gonadotropin dosage and an association between serum FSH (follicular stimulating hormone) levels during stimulation and response will be assessed.
  Blood samples will be taken (along with clinical standard routine) on day 2/3 of cycle, day 5 / 8 and 10 of stimulation and on the day of trigger (DoT). Urine samples will be taken additionally.
  Final oocyte maturation will be triggered with 250 mcg recombinant human Choriogonadotropin and 0.2 mg Decapeptyl as soon as >2 follicles reach 17 mm diameter.
  Women who have more than 30 follicles ≥12 mm and or serum estradiol levels above>5000 pg/ml on the day of trigger will only be triggered with Decapeptyl. OPU (oocyte pick up) will be 36 h after trigger.
  On the day of oocyte collection (OPU), follicular fluid from the largest follicle will be checked for FSH level after the cumulus oocyte complex is removed.
  Interventions: Drug: Gonal-f (gonadotropin)

INTERVENTIONS:
Drug: Gonal-f (gonadotropin) — Women will be given 300 IU Gonal-F daily from cycle day 2 or 3. Gonal F will be injected at 8 pm daily. They will all receive cetrorelix acetate 250 mcg/day (Cetrotide) subcutaneously from stimulation day 5 onwards until and including the trigger day. Cetrotide will be administered at 08:00 am.

SUMMARY:
This study examines if monitoring serum Follicle Stimulation Hormone (FSH) levels can predict oocyte yield and progesterone levels, considering factors like age, baseline FSH, Antral Mullerian Hormone (AMH), antral follicle count, body weight, kidney function, and urinary FSH. The aim is to find a minimum FSH level that ensures optimal ovarian response and enables tailored FSH dosages for better outcomes.

DETAILED DESCRIPTION:
Ovarian stimulation typically uses transvaginal ultrasound to monitor follicle growth and endometrial condition, with some clinics also tracking serum estradiol and progesterone levels, but often neglecting serum Follicle Stimulation Hormone (FSH). FSH is essential for follicle development, yet its levels can vary widely among women receiving the same dose due to factors like body weight, renal function, and ovarian reserve.

This study aims to identify a minimum effective FSH threshold that ensures optimal follicular growth while avoiding excess administration.

ELIGIBILITY:
Inclusion Criteria:

* regular 21 - 35 days cycles
* BMI between 19 - 30 kg/m2
* serum AMH level between 1.5 to 3 ng/ml
* a total antral follicle count between 10 to 24
* endogenous early follicular phase serum FSH level <10 IU/L
* normal glomerular filtration rate

Exclusion Criteria:

* hypogonadotropic hypogonadism
* history of ovarian surgery
* permanent ovarian cysts of any form
* older than 39 years
* abnormal thyroid stimulating hormone (TSH)
* renal disease
* elevated prolactin levels
* intake of oral contraceptives 3 months before stimulation start and estradiol pretreatment will be excluded

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between 18 and 39 years old, with regular 21 - 35 days cycles, BMI between 19 - 30 kg/m2, serum AMH level between 1.5 to 3 ng/ml, a total antral follicle count between 10 to 24, endogenous early follicular phase serum FSH level <10 IU/L, normal glomerular filtration rate who is planned to undergo ovarian stimulation in a Gonadotropin hormone-releasing hormone (GnRH) antagonist protocol can be included.
  Exclusion will be for women with hypogonadotropic hypogonadism, history of ovarian surgery, permanent ovarian cysts of any form, older than 39 years, abnormal thyroid function (TSH level outside the normal range), renal disease, elevated prolactin levels. intake of oral contraceptives 3 months before stimulation start and estradiol pretreatment will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative Measurement of Serum Follicle-Stimulating Hormone (FSH) Levels During Ovarian Stimulation Using Serum Assays. | 1 year
  serum FSH levels during ovarian stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- ART Fertility Clinics, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
on request

REFERENCES:
- [Background] Filicori M, Cognigni GE, Gamberini E, Parmegiani L, Troilo E, Roset B. Efficacy of low-dose human chorionic gonadotropin alone to complete controlled ovarian stimulation. Fertil Steril. 2005 Aug;84(2):394-401. doi: 10.1016/j.fertnstert.2005.02.036. PMID 16084880
- [Background] Huber M, Hadziosmanovic N, Berglund L, Holte J. Using the ovarian sensitivity index to define poor, normal, and high response after controlled ovarian hyperstimulation in the long gonadotropin-releasing hormone-agonist protocol: suggestions for a new principle to solve an old problem. Fertil Steril. 2013 Nov;100(5):1270-6. doi: 10.1016/j.fertnstert.2013.06.049. Epub 2013 Aug 6. PMID 23931964
- [Background] Jeppesen JV, Kristensen SG, Nielsen ME, Humaidan P, Dal Canto M, Fadini R, Schmidt KT, Ernst E, Yding Andersen C. LH-receptor gene expression in human granulosa and cumulus cells from antral and preovulatory follicles. J Clin Endocrinol Metab. 2012 Aug;97(8):E1524-31. doi: 10.1210/jc.2012-1427. Epub 2012 Jun 1. PMID 22659248
- [Background] La Marca A, Sunkara SK. Individualization of controlled ovarian stimulation in IVF using ovarian reserve markers: from theory to practice. Hum Reprod Update. 2014 Jan-Feb;20(1):124-40. doi: 10.1093/humupd/dmt037. Epub 2013 Sep 29. PMID 24077980
- [Background] Lawrenz B, Melado L, Digma S, Sibal J, Coughlan C, Andersen CY, Fatemi HM. Reintroducing serum FSH measurement during ovarian stimulation for ART. Reprod Biomed Online. 2022 Mar;44(3):548-556. doi: 10.1016/j.rbmo.2021.10.020. Epub 2021 Oct 31. PMID 34973935
- [Background] Macklon NS, Stouffer RL, Giudice LC, Fauser BC. The science behind 25 years of ovarian stimulation for in vitro fertilization. Endocr Rev. 2006 Apr;27(2):170-207. doi: 10.1210/er.2005-0015. Epub 2006 Jan 24. PMID 16434510